CLINICAL TRIAL: NCT03050437
Title: A Randomized, Open Label, Phase II Study Comparing Pemetrexed Plus Cisplatin Followed by Pemetrexed Until Progression Versus Pemetrexed Alone Until Progression in Non-small Cell Lung Cancer Patients Who Have Progressed on First Line Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI)
Brief Title: A Study Comparing Pemetrexed Plus Cisplatin Versus Pemetrexed Alone in NSCLC Patients Who Have Progressed on First Line EGFR-TKI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-12-035
Record Dates: First submitted 2015-09-22; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Failed in First Line EGFR-TKI; EGFR Activating Mutation; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pem/Cis (Experimental): Pem/Cis IV every 3 weeks
  Interventions: Drug: Cisplatin; Drug: Pemetrexed
- Pem alone (Active Comparator): Pem IV alone every 3 weeks
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Cisplatin — cisplatin is added to Pem/cis arm
  Arms: Pem/Cis
Drug: Pemetrexed — Pem is applied to both arms

SUMMARY:
It has not been established whether platinum-based doublets is better than single agent chemotherapy in EGFR mutant NSCLC patients who failed first-line EGFR TKI.

In this prospective trial, the investigators try to evaluate whether the progression-free survival of pemetrexed/cisplatin (PC) regimen is longer than that of pemetrexed single(P) regimen in NSCLC patients who have progressed after first line treatment of EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nonsquamous NSCLC with activating EGFR mutation (on exon 19 deletion or exon 21 L858R mutation)
* Stage IIIb, IV or recurrent NSCLC (AJCC 7th criteria)
* Age ≥ 20 years
* ECOG performance status of 0 or 1
* At least one measurable lesion by RECIST 1.1
* Progression after first line treatment with EGFR TKIs for advanced NSCLC
* Asymptomatic brain metastasis or symptomatic brain metastasis treated with local treatment such as operation, whole brain radiotherapy, or gamma-knife surgery
* At least 2 weeks later after whole brain radiotherapy or palliative radiotherapy
* Adequate renal function: estimated creatinine clearance ≥ 45 mL/min
* Organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 3 UNL, in case of known hepatic metastasis, AST/ALT< 5 UNL
* Written informed consent form
* No other previous systemic chemotherapy

Exclusion Criteria:

* Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
* Patients with post-obstructive pneumonia or uncontrolled serious infection
* Pregnant or nursing women (Women of reproductive potential have to agree to use an effective contraceptive method)
* Uncontrolled symptomatic brain metastasis
* Presence of third space fluid which cannot be controlled by drainage
* Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea